CLINICAL TRIAL: NCT00524966
Title: Randomized Controlled Trial of Bipolar Versus Ultrasonic Hemostasis Techniques in Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Electron Kebebew, MD, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Harmonic
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-07

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Second Harmonic Generation Microscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Bipolar Versus Ultrasonic Hemostasis Techniques — OUTLINE: Patients undergoing thyroidectomy for thyroid cancer, thyroid nodules, hyperthyroidism and goiter will be randomized to either bipolar energy sealing system or ultrasonic coagulation.
  Other Names: Harmonic; LigaSure

SUMMARY:
RATIONALE: The use of bipolar energy sealing system or ultrasonic coagulation for hemostasis during thyroidectomy may reduce blood loss and hypocalcemia and may be more cost-effective.

DETAILED DESCRIPTION:
PURPOSE: This clinical trial is studying how well bipolar energy sealing system and ultrasonic coagulation for hemostasis during thyroidectomy reduce blood loss and hypocalcemia, as well as which device is the most cost-effective approach for thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring thyroidectomy

Exclusion Criteria:

* Patients unwilling or unable to provide informed consent
* Age less than 18 years old
* Reoperative case
* Patients who use pacemakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Blood loss and hypocalcemia | one week

SECONDARY OUTCOMES:
Cost of thyroidectomy | one week

CONTACTS AND LOCATIONS:
Overall Officials: Electron Kebebew, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Comprehensive Cancer Center, San Francisco, California, United States